CLINICAL TRIAL: NCT00006327
Title: A Phase III Trial to Determine the Efficacy of AIDSVAX B/E Vaccine in Intravenous Drug Users in Bangkok, Thailand
Brief Title: Effectiveness of AIDSVAX B/E Vaccine in Intravenous Drug Users in Bangkok, Thailand
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VaxGen (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Prevention
Other Study IDs: VAX 003
Record Dates: First submitted 2000-10-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-06

CONDITIONS: HIV Infections; HIV Seronegativity
Keywords: Recombinant Proteins; HIV-1; AIDS Serodiagnosis; Substance Abuse, Intravenous; Enzyme-Linked Immunosorbent Assay; Blotting, Western; HIV Envelope Protein gp120; AIDSVAX
MeSH Terms: conditions — HIV Infections; Substance Abuse, Intravenous

INTERVENTIONS:
Biological: MN rgp120/HIV-1 and A244 rgp120/HIV-1

SUMMARY:
The purpose of this study is to determine if the vaccine, AIDSVAX B/E, will protect intravenous drug users from becoming infected with HIV.

DETAILED DESCRIPTION:
Volunteers are immunized and followed for a minimum of 2 years. Any volunteer that becomes infected with HIV-1 is followed every 4 months post infection for up to 36 months. Behavior effects associated with study participation are assessed.

ELIGIBILITY:
Inclusion Criteria

Volunteers may be eligible for this study if they:

* Are 20 to 60 years old.
* Are HIV-negative.
* Have used intravenous drugs in the previous 12 months.
* Are available and commit to 3 years of follow-up.
* Have a Thai National ID or its equivalent such as government official ID or state enterprise ID.
* Are able to understand the study and pass a test showing they understand it, and give written informed consent.

Exclusion Criteria

Volunteers will not be eligible for this study if they:

* Have a serious disease or condition, or history of a serious disease or condition such as lymphoma, that would interfere with the study.
* Are HIV-positive.
* Have ever received an experimental HIV-1 vaccine.
* Have had or expect to have any treatments or medications that interfere with the immune system (e.g., long-term use of systemic steroids, chemotherapy, or radiation).
* Have received a vaccine or immunoglobulin within 2 weeks of receiving the first study injection, or other vaccines within 4 weeks of the first study injection.
* Have received immunoglobulins for a long time.
* Have received non-licensed, research agents within 4 weeks of the first study injection.
* Expect to miss study visits or plan to move within 36 months.
* Are pregnant or breast-feeding or plan to become pregnant during the 36-month study period.
* Are women who have sex with men and do not plan to use effective birth control.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2500
Dates: Start 1999-03; Study Completion 2000-08

CONTACTS AND LOCATIONS:
Overall Officials: Kachit Choopanya, Principal Investigator
Locations (1):
- Kachit Choopanya, Klongsan / Bangkok, Thailand

REFERENCES:
- [Derived] Martin M, Vanichseni S, Suntharasamai P, Mock PA, van Griensven F, Pitisuttithum P, Tappero JW, Chiamwongpaet S, Sangkum U, Kitayaporn D, Gurwith M, Choopanya K; Bangkok Vaccine Evaluation Group. Drug use and the risk of HIV infection amongst injection drug users participating in an HIV vaccine trial in Bangkok, 1999-2003. Int J Drug Policy. 2010 Jul;21(4):296-301. doi: 10.1016/j.drugpo.2009.12.002. Epub 2010 Jan 15. PMID 20079620
- [Derived] Suntharasamai P, Martin M, Vanichseni S, van Griensven F, Mock PA, Pitisuttithum P, Tappero JW, Sangkum U, Kitayaporn D, Gurwith M, Choopanya K; Bangkok Vaccine Evaluation Group. Factors associated with incarceration and incident human immunodeficiency virus (HIV) infection among injection drug users participating in an HIV vaccine trial in Bangkok, Thailand, 1999-2003. Addiction. 2009 Feb;104(2):235-42. doi: 10.1111/j.1360-0443.2008.02436.x. PMID 19149819